CLINICAL TRIAL: NCT01065324
Title: Intestinal Barrier Permeability Defects, Recovery, and Risk of Bacterial Translocation Induced After Deep Intestinal Manipulation by Balloon-assisted Enteroscopy: From Basic to Clinical Research
Brief Title: Balloon-assisted Enteroscopy and Bacteria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: NTUH, NTUH
Other Study IDs: 200812154R
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Enteritis; Bleeding
Keywords: balloon; enteroscopy; bacteremia
MeSH Terms: conditions — Enteritis; Hemorrhage; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial DNA, host DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anally inserted enteroscopy group: Anally inserted enteroscopy group
- Orally inserted enteroscopy group: Orally inserted enteroscopy group

SUMMARY:
1. Balloon-assisted enteroscopy (BAE) is a new tool to investigate small intestinal diseases.
2. Deep enteroscopy made possible by balloon expansion and manipulation of small intestines.
3. However, whether intestinal barrier injured during BAE predispose patients to bacteremia or clinical relevant infection is not studied.
4. We will also examine relevant patient factors.

DETAILED DESCRIPTION:
The newly developed balloon-assisted enteroscopy systems allow insertion of the enteroscopy deeply into the small intestines by fixation of the soft, redundant small intestines with an inflatable balloon over the tip of the overtube. However, the inflation of balloon might stimulate the intestinal mucosa, and the deep manipulation of intestinal segments might also compromise the intestinal barrier function. According to our preliminary experience of balloon-assisted enteroscopy (which is among the first groups in Taiwan), we experienced a significant case of suspected post-procedural bactermia patient. Besides, there is also a published case report from the UK reporting Streptococcus milleri bacteremia which is suspected as bacterial translocation after balloon-assisted enteroscopy. However, currently there is no original study focusing on the intestinal barrier / permeability defects or bacterial translocation. This is a timely and novel research topic in the current developing era of balloon-assisted enteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with clinical suspicions of small intestinal lesions in need of balloon-assisted enteroscopy examinations
* signed written informed consents

Exclusion Criteria:

* Patients with active infection or receiving systemic (oral or intravenous) antibiotics within recent 3 months (this may decrease effect of bacterial translocation) or taking drugs that may affect renal function within 3 months
* Unstable health condition for balloon-assisted enteroscopy (unstable hemodynamics, severe cardiopulmonary compromise)
* Pregnancy
* known allergy to lactulose, mannitol
* Refuse to sign written informed consent of this study.
* patients would be advised to hold prokinetic agents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary medical center,patients with clinical presentation necessitating deep enteroscopy examinations.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-02; Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
molecular bacteremia | 7d

CONTACTS AND LOCATIONS:
Overall Officials: TC Lee, MD, Principal Investigator — NTUH
Locations (2):
- Taiwan (2):
  - E-Da Hospital, Kaohsiung City
  - NTUH, Taipei